CLINICAL TRIAL: NCT03955536
Title: Comparison of the Effects of Different Physiotherapy and Rehabilitation Methods in Phase I Following Open Heart Surgery
Brief Title: Comparison of the Effects of Different Physiotherapy and Rehabilitation Methods on Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Beykent (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Lecturer, University of Beykent
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UBeykent
Record Dates: First submitted 2019-03-22; First posted 2019-05-20 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Open Heart Surgery
Keywords: Cardiac Rehabilitation; Virtual Reality; Respiratory Muscle Training; Open Heart Surgery

STUDY DESIGN:
Intervention Model Description: randomized controlled trial 3 groups
  1. Group routine cardiac rehabilitation program (RCRP)
  2. Group RCRP and inspiratory muscle training
  3. Group RCRP and virtual reality application
Who Masked: Participant
Masking Description: Inclusion criteria 25-70 age range Undergoing open heart surgery Hemodynamically stable Ambulatory No advanced vision defect The physician authorized by the operating physician for participation in the exercise Patients who agreed to participate in the study. Exclusion criteria The presence of pulmonary, neurological, musculoskeletal disease limiting participation in exercise training Patients at high risk (ejection fraction below 40 percent) Dissectant aneurysm Patients who cannot be cooperative in verbal and / or auditory terms Psychological and / or perceptual cooperative patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Routine cardiac rehabilitation program (RCRP)atient education
  Interventions: Other: Group A: Group routine cardiac rehabilitation program (RCRP)
- Group B (Experimental): routine cardiac rehabilitation program + virtual reality
  Interventions: Other: Group B: Group RCRP and inspiratory muscle training
- Group C (Experimental): RCRP + inspiratory muscle training
  Interventions: Other: Group C: Group RCRP and virtual reality application

INTERVENTIONS:
Other: Group A: Group routine cardiac rehabilitation program (RCRP) — Patient education, Chest Physiotherapy, Abdominal and chest breathing, Bronchial hygiene techniques, Segmental breathing exercises, Triflow, exercise and mobilization,graduated exercise, positioning, active joint movement, moving inside bed, sitting at the edge of the bed, transfer from bed to chair, standing walking program, up and down stairs.
  Evaluations for each patient (preoperative and just before discharge) Spirometric measurements Intraoral pressure measurementDyspnea assessment (BORG), Pain assessment (VAS), Evaluation of anxiety and depression (HAD) Evaluation of functional capacity (6 minutes walking test) Quality of Life (MacNew Heart Disease Specific Quality of Life Questionnaire)
  Arms: Group A
Other: Group B: Group RCRP and inspiratory muscle training — use of additional virtual reality goggles in the routine cardiac rehabilitation program Virtual reality glasses installed in the patient will feel the best way to feel an environment.
  Virtual reality glasses are planned to be used 15 minutes by increasing the usage period.
  Evaluations for each patient (preoperative and just before discharge) Spirometric measurements Intraoral pressure measurementDyspnea assessment (BORG), Pain assessment (VAS), Evaluation of anxiety and depression (HAD) Evaluation of functional capacity (6 minutes walking test) Quality of Life (MacNew Heart Disease Specific Quality of Life Questionnaire)
  Arms: Group B
Other: Group C: Group RCRP and virtual reality application — nspiratory muscle training with "Threshold" for routine cardiac rehabilitation Training intensity
  - 30% of the maximum measured inspiratory pressure per week (15 min.). Every 10 breaths after rest.
  Evaluations for each patient (preoperative and just before discharge) Spirometric measurements Intraoral pressure measurementDyspnea assessment (BORG), Pain assessment (VAS), Evaluation of anxiety and depression (HAD) Evaluation of functional capacity (6 minutes walking test) Quality of Life (MacNew Heart Disease Specific Quality of Life Questionnaire)
  Arms: Group C

SUMMARY:
The aim of this study is to compare the effects of different physiotherapy and rehabilitation methods in hospitalization after Open Heart Surgery (OHS). In this context, it is planned that patients undergoing OHS surgery will be randomly divided into 3 groups.

1. Group routine cardiac rehabilitation program (RCRP)
2. Group RCRP and inspiratory muscle training
3. Group RCRP and virtual reality application Treatment of patients will be administered twice daily during their stay in the hospital. The patients will be evaluated by clinical measurements and scales based on patient notification and before and after the treatment and their effectiveness and superiority over each other will be determined.

DETAILED DESCRIPTION:
Purpose of our study Comparison of the effects of different physiotherapy and rehabilitation methods in hospitalization after Open Heart Surgery (OHS).

Expected results: Routine cardiac rehabilitation program (RCRP) + virtual reality group and RCRP + inspiratory muscle training group pain, dyspnea, anxiety, depression, quality of life, respiratory muscle strength We believe that there will be good progress in pulmonary function, 6 minutes walking distance evaluation results, and best developments will occur in RCRP + virtual reality + inspiratory muscle training group.

In this context, it is planned that patients undergoing OHS surgery will be randomly divided into 3 groups. Group 1 routine cardiac rehabilitation program (RCRP) 2. Group RCRP and inspiratory muscle training 3. Group RCRP and virtual reality application Treatment of patients will be administered twice daily during their stay in the hospital. The patients will be evaluated by clinical measurements and scales based on patient notification and before and after the treatment and their effectiveness and superiority over each other will be determined.

Literature summary:

Open Heart Surgery is one of the most effective and reliable treatment options in coronary artery diseases and the most common coronary artery bypass surgery in the world is used to prolong the life expectancy of patients and reduce symptoms. Patients undergoing cardiac rehabilitation program after Open Heart Surgery are extremely important and the benefits of cardiac rehabilitation; reduction in symptoms, exercise tolerance and increase in workforce, improvement in blood lipid and general risk profile, decrease in smoking, stress management and self-improvement, atherosclerotic status, new coronary attacks, hospitalizations, decreases in morbidity and mortality.Despite the well-known positive effects of open heart surgery, respiratory complications are common in patients with decreased respiratory muscle strength in the postoperative period.

Inspiratory muscle training with yararlı Threshold iştir performed after open heart surgery helps to increase respiratory muscle strength and endurance, and potential beneficial effects have been demonstrated in cardiac patients undergoing coronary artery bypass surgery.

In a randomized controlled trial of 38 patients undergoing coronary artery bypass surgery, respiratory muscle training has been shown to provide improvements in maximum inspiratory pressure, maximum expiratory pressure, peak flow rate, and tidal volume results. In another randomized controlled trial of 47 patients with coronary artery bypass surgery, the patients' postoperative ventilation capacity and respiratory muscle strength decreased. It was reported that inspiratory muscle training increased the tidal volume and vital capacity parameters.

Hospitalization is an experience that increases the anxiety and anxiety of the individual. Individual in the hospital environment; they may feel threatened, feel fear and insecurity. Using virtual reality glasses can help patients to feel different in a different environment. This may be beneficial to the patient in eliminating the negative emotions brought by the hospital environment and may positively affect their participation in the treatment.

Virtual reality applications, which have gained importance in many areas of medicine, have shown that improved exercise programs and enriched environment provide better functional performance in patients undergoing cardiac surgery. After reviewing the literature related to virtual reality combined rehabilitation applications after coronary artery bypass surgery, there are only three studies in the form of walking and exercise training in virtual environment.

In a randomized controlled trial of 60 patients undergoing coronary artery bypass surgery, the patients were divided into two groups: the traditional cardiac rehabilitation group and the additional virtual reality group of traditional cardiac rehabilitation. The patients were evaluated on the day of preoperative, postoperative first, third and discharge days with Functional Independence Measurement (FIM), 6 Minute Walk Test and Nottigham Health Profile. Traditional cardiac rehabilitation program applied to both groups twice a day was determined as breathing exercises, airway cleaning techniques, metabolic and motor exercise training. In the study group, motor exercises in traditional cardiac rehabilitation program were performed twice a day using virtual reality and kinesiotherapy. As a result of evaluations, cardiac rehabilitation combined with virtual reality application has been shown to provide better functional performance in patients.

In 2006, 20 patients who had undergone coronary artery bypass surgery were included. It has been shown that a rehabilitation program with virtual reality applications is useful to improve the physical capacity of patients. In another study conducted on 32 patients undergoing coronary artery bypass surgery in 2005, it was reported that the inclusion of a virtual reality environment in cardiac rehabilitation programs would accelerate the maximum recovery of patients' cardiovascular functions.

In the literature, there is no study in which the inspiratory muscle training was performed in a virtual environment created by virtual reality glasses.

ELIGIBILITY:
Inclusion Criteria:

* 25-70 age range
* Undergoing open heart surgery
* Hemodynamically stable
* Ambulatory
* No advanced vision defect
* The physician authorized by the operating physician for participation in the exercise
* Patients who agreed to participate in the study.

Exclusion Criteria:

* The presence of pulmonary, neurological, musculoskeletal disease limiting participation in exercise training
* Patients at high risk (ejection fraction below 40 percent)
* Dissectant aneurysm
* Patients who cannot be cooperative in verbal and / or auditory terms
* Psychological and / or perceptual cooperative patients

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of respiratory functions with simple spirometric measurements | the preoperative and 10th day
  spirometric measurement with spirometry
intraoral pressure measurement (Maximum inspiratory pressure maximum expiratory pressure) | the preoperative and 10th day
  Maximum inspiratory pressure maximum expiratory pressure

SECONDARY OUTCOMES:
Dyspnea assessment | the preoperative and 10th day
  With modified borg dyspnea scale:
  Modified Borg Scale is a scale that is frequently used to evaluate the intensity of dyspnea and the severity of rest dyspnea. It consists of ten items that define the severity of dyspnea according to their degree. The high score is directly proportional to the severity of dyspnea.
Peak expiratory flow | the preoperative and 10th day
  peak flow meter
Evaluation of functional capacity with 6 minutes walking test | the preoperative and 10th day
  With 6 minutes walking test:
  The 6-minute walk test is one of the functional exercise capacity assessment tests. In this test, participants are asked to walk as long as possible within 6 minutes in a 30 meter (m) corridor. When they feel fatigue or pain, they are advised to stop and rest when they feel ready to walk. At the end of 6 minutes, the total distance of the patients walking is recorded. Heart rates, systolic and diastolic blood pressures, O2 saturation, perceived fatigue and dyspnea levels are recorded before and after the test.
Evaluation of anxiety and depression | the preoperative and 10th day
  With hospital anxiety and depression scale(HAD):
  The HADS includes anxiety and depression subscales. The scale is a self-report scale and consists of 14 items, 7 of which are depression (even numbers) and 7 are anxiety symptoms (odd numbers).
Pain assessment | the preoperative and 10th day
  With Visuel Analog Scale:
  Participants are asked to mark the point where they feel their pain on a 10 centimeter (cm) horizontal line. 0-no pain, 10-unbearable pain. Night, activity and pain conditions are evaluated separately at rest.
Quality of Life assessment | the preoperative and 10th day
  MacNew Heart Disease Specific Quality of Life Questionnaire:
  The Mac New Heart Disease Quality of Life Questionnaire is designed to assess how patients' physical, emotional, social functions and daily activities are affected over a 2-week period. The scale consists of three sub-dimensions and 27 items, some of which are into more than one sub-dimension. The subscale scores are calculated by taking the environments of the responses to the questions in each sub-dimension, and when the possible scores vary between 1-7, the higher scores indicate a better quality of life. The Turkish validity and reliability study of the scale was performed in 2008 by Daskapan et al. made by.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Şahbaz, Principal Investigator — researcher
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Alexander JH, Smith PK. Coronary-Artery Bypass Grafting. N Engl J Med. 2016 May 19;374(20):1954-64. doi: 10.1056/NEJMra1406944. No abstract available. PMID 27192673
- [Background] Barros GF, Santos Cda S, Granado FB, Costa PT, Limaco RP, Gardenghi G. Respiratory muscle training in patients submitted to coronary arterial bypass graft. Rev Bras Cir Cardiovasc. 2010 Oct-Dec;25(4):483-90. doi: 10.1590/s0102-76382010000400011. English, Portuguese. PMID 21340377
- [Background] Cacau Lde A, Oliveira GU, Maynard LG, Araujo Filho AA, Silva WM Jr, Cerqueria Neto ML, Antoniolli AR, Santana-Filho VJ. The use of the virtual reality as intervention tool in the postoperative of cardiac surgery. Rev Bras Cir Cardiovasc. 2013 Jun;28(2):281-9. doi: 10.5935/1678-9741.20130039. PMID 23939326
- [Background] Chuang TY, Sung WH, Chang HA, Wang RY. Effect of a virtual reality-enhanced exercise protocol after coronary artery bypass grafting. Phys Ther. 2006 Oct;86(10):1369-77. doi: 10.2522/ptj.20050335. PMID 17012641
- [Background] Chuang TY, Sung WH, Lin CY. Application of a virtual reality-enhanced exercise protocol in patients after coronary bypass. Arch Phys Med Rehabil. 2005 Oct;86(10):1929-32. doi: 10.1016/j.apmr.2005.05.003. PMID 16213233
- [Background] Ferreira PE, Rodrigues AJ, Evora PR. Effects of an inspiratory muscle rehabilitation program in the postoperative period of cardiac surgery. Arq Bras Cardiol. 2009 Apr;92(4):275-82. doi: 10.1590/s0066-782x2009000400005. English, Portuguese, Spanish. PMID 19565135
- [Background] Ghoneim MM, O'Hara MW. Depression and postoperative complications: an overview. BMC Surg. 2016 Feb 2;16:5. doi: 10.1186/s12893-016-0120-y. PMID 26830195
- [Background] Gomes Neto M, Martinez BP, Reis HF, Carvalho VO. Pre- and postoperative inspiratory muscle training in patients undergoing cardiac surgery: systematic review and meta-analysis. Clin Rehabil. 2017 Apr;31(4):454-464. doi: 10.1177/0269215516648754. Epub 2016 Jul 10. PMID 27154820
- [Background] Herdy AH, Marcchi PL, Vila A, Tavares C, Collaco J, Niebauer J, Ribeiro JP. Pre- and postoperative cardiopulmonary rehabilitation in hospitalized patients undergoing coronary artery bypass surgery: a randomized controlled trial. Am J Phys Med Rehabil. 2008 Sep;87(9):714-9. doi: 10.1097/PHM.0b013e3181839152. PMID 18716482
- [Background] Matheus GB, Dragosavac D, Trevisan P, Costa CE, Lopes MM, Ribeiro GC. Inspiratory muscle training improves tidal volume and vital capacity after CABG surgery. Rev Bras Cir Cardiovasc. 2012 Jul-Sep;27(3):362-9. doi: 10.5935/1678-9741.20120063. English, Portuguese. PMID 23288176
- [Background] Poole L, Kidd T, Leigh E, Ronaldson A, Jahangiri M, Steptoe A. Psychological distress and intensive care unit stay after cardiac surgery: The role of illness concern. Health Psychol. 2015 Mar;34(3):283-7. doi: 10.1037/hea0000183. Epub 2014 Dec 22. PMID 25528184
- [Background] Spiroski D, Andjic M, Stojanovic OI, Lazovic M, Dikic AD, Ostojic M, Beleslin B, Kostic S, Zdravkovic M, Lovic D. Very short/short-term benefit of inpatient/outpatient cardiac rehabilitation programs after coronary artery bypass grafting surgery. Clin Cardiol. 2017 May;40(5):281-286. doi: 10.1002/clc.22656. Epub 2017 Jan 11. PMID 28075500
- [Background] Valkenet K, de Heer F, Backx FJ, Trappenburg JC, Hulzebos EH, Kwant S, van Herwerden LA, van de Port IG. Effect of inspiratory muscle training before cardiac surgery in routine care. Phys Ther. 2013 May;93(5):611-9. doi: 10.2522/ptj.20110475. Epub 2013 Jan 3. PMID 23288909